CLINICAL TRIAL: NCT04945096
Title: Outcomes of Patients After Allogenic Hematopoietic Cell Transplantation With Decitabine-containing Conditioning Regimen and Acetylcysteine Treatment
Brief Title: Outcomes of Patients After Allo-HSCT With Decitabine and NAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2021-1
Record Dates: First submitted 2021-04-25; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-04

CONDITIONS: Engraft Failure; Relapse; GVHD
MeSH Terms: conditions — Recurrence | interventions — Decitabine; Acetylcysteine; Semustine; Cytarabine; Busulfan; Cyclophosphamide; Cyclosporine; Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized after the investigator has verified that all eligibility criteria have been met. Subjects will be randomized in a 1:1 ratio to either Experimental Group (Acetylcysteine + Decitabine) or Active Comparator Group (Standard Treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetylcysteine + decitabine (Experimental): Acetylcysteine (1.2g twice a day, oral administration, from day -10 to day 365 after HSCT). Conditional regimen: decitabine (20mg/m2 intravenously from day -10 to day -8 of conditional regimen); semustine 250 mg/m2/day on day -9; cytarabine 2 g/m2 every 12 hours on day -8; busulfan 3.2mg/kg/day on day -7 to -5; cyclophosphamide 1.8g/m2/day on day -4 to -3; cyclosporin A: 3mg/kg/d from day -8. Anti-thymocyte globulin (2mg/kg/d on day -5 to day -2) and mycophenolate (500mg, oral, twice a day from day -8) were usually added for transplants with unrelated donor or HLA mismatched donor.
  Interventions: Drug: decitabine; Drug: Acetylcysteine; Drug: Semustine; Drug: Cytarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporin A; Drug: Anti-thymocyte globulin; Drug: Mycophenolate
- Standard Treatment (Active Comparator): Conditional regimen: semustine 250 mg/m2/day on day -9; cytarabine 2 g/m2 every 12 hours on day -8; busulfan 3.2mg/kg/day on day -7 to -5; cyclophosphamide 1.8g/m2/day on day -4 to -3; cyclosporin A: 3mg/kg/d from day -8. Anti-thymocyte globulin (2mg/kg/d on day -5 to day -2) and mycophenolate (500mg, oral, twice a day from day -8) were usually added for transplants with unrelated donor or HLA mismatched donor.
  Interventions: Drug: Semustine; Drug: Cytarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporin A; Drug: Anti-thymocyte globulin; Drug: Mycophenolate

INTERVENTIONS:
Drug: decitabine — Decitabine (20mg/m2 intravenously from day -10 to day -8 of conditional regimen)
  Other Names: 5-aza-2'-deoxycytidine
  Arms: Acetylcysteine + decitabine
Drug: Acetylcysteine — Acetylcysteine: 1.2g twice a day, oral administration, from day -10 to day 365 after HSCT.
  Other Names: Acetadote
  Arms: Acetylcysteine + decitabine
Drug: Semustine — Semustine: 250 mg/m2/day on day -9.
  Other Names: Methyl-CCNU
Drug: Cytarabine — Cytarabine: 2 g/m2 every 12 hours on day -8.
  Other Names: Cytosine arabinoside
Drug: Busulfan — Busulfan: 3.2mg/kg/day on day -7 to -5.
  Other Names: Myleran
Drug: Cyclophosphamide — Cyclophosphamide: 1.8g/m2/day on day -4 to -3.
  Other Names: Cytoxan
Drug: Cyclosporin A — Cyclosporin A: 3mg/kg/d from day -8.
  Other Names: Cyclosporine
Drug: Anti-thymocyte globulin — Anti-thymocyte globulin (2mg/kg/d on day -5 to day -2) will be added for transplants with unrelated donor or HLA mismatched donor.
  Other Names: Thymoglobulin
Drug: Mycophenolate — Mycophenolate (500mg, oral, twice a day from day -8) will be added for transplants with unrelated donor or HLA mismatched donor.
  Other Names: CellCept

SUMMARY:
The investigators will conduct this prospective and randomized clinical trial, to evaluate the hematopoietic reconstitution, GVHD and relapse rate of patients after allo-HSCT with decitabine containing conditional regimen and NAC treatment.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the main curative treatment for hematological malignancy. Relapse, graft versus host disease (GVHD) and graft failure are the main causes of treatment failure. Acetylcysteine (NAC) was found to be able to enhance defective HSCs by repairing dysfunctional bone marrow endothelial cells, and overcome the exhaustion of HSCs and enhance the engraftment of HSCs. Decitabine could restore bone marrow microenvironment by repairing endothelial cells and endothelial progenitor cells, as well as cytokines and chemokines which are crucial to HSCs proliferation and differentiation, thereby promote platelet recovery after HSCT. Besides, decitabine therapy was shown to be associated with reduced incidence of GVHD, lower relapse rate, and increased overall survival in several studies. Thereby the investigators will conduct this clinical trial to evaluate the hematopoietic reconstitution, GVHD and relapse rate of patients with hematological malignancy after allo-HSCT with decitabine containing conditional regimen and NAC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as hematopoietic malignancy;
2. Achieved complete remission since the last chemotherapy;
3. Age 10-70 years；
4. Be willing to receive allo-HSCT, with HLA matched related or HLA matched unrelated, or HLA mismatched related donor.

Exclusion Criteria:

1. Active infections, severe organ damage (cardiac, renal and/or hepatic dysfunction greater than grade 2 according to the Common Terminology Criteria for Adverse Events V5.0), or any other conditions that make patients ineligible for allo-HSCT;
2. Allergic to acetylcysteine or decitabine.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The hematological engraftment rates | 1 year
  The hematological engraftment rates of patients after HSCT.
GVHD rates | 1 year
  The GVHD rates of patients after HSCT.
Relapse rates | 1 year
  The relapse rates of patients after HSCT.

SECONDARY OUTCOMES:
Overall survival | 1 year
  To evaluate the overall survival (days) of patients after HSCT.
Disease free survival | 1 year
  To evaluate the disease free survival (days) of patients after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Prof., Study Chair — The First Affiliated Hospital of Soochow University

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT04945096/Prot_SAP_ICF_000.pdf